CLINICAL TRIAL: NCT00246818
Title: A Randomized Study of the Effect of Tai Chi Chuan Compared to a Structured Exercise Program on Parameters of Physical Fitness and Stress in Adult Cancer Survivors
Brief Title: Effect of Tai Chi Vs. Structured Exercise on Physical Fitness and Stress in Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060016; 06-AT-0016; NCT00414791 (obsolete NCT alias)
Record Dates: First submitted 2005-10-29; First posted 2005-10-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-25

CONDITIONS: Cancer; Cancer Survivor
Keywords: Mind-Body; Stress Reduction; Complementary Medicine; Quality of Life; Well-being; Psychoneuroimmunology; Tai Chi; Aerobic Exercise; Cancer Survivor
MeSH Terms: conditions — Neoplasms | interventions — Tai Ji

INTERVENTIONS:
Procedure: Tai Chi Chuan

SUMMARY:
This study will compare the effectiveness of Tai Chi (a sequence of slow, graceful body movements) and a cardiovascular exercise fitness program in improving physical fitness and endurance, reducing stress and improving well-being in adult survivors of cancer. Tai Chi, described by some as a moving form of yoga and meditation combined, evolved from martial arts and breathing exercises in China hundreds of years ago. This study uses the 24-posture standardized Tai Chi. The movements are continuous, smooth, and natural, with the upper and lower parts of the body following each other. The entire body is always in motion, with the movements performed gently and at a uniform speed. The exercise training program uses an exercise machine. The training regimen is adjusted to maintain the individual's average training heart rate at 70 to 80 percent heart rate reserve; i.e., 220 minus the person's age.

Cancer survivors of solid tumor cancers who are between 18 and 65 years of age, whose treatment included chemotherapy, biologic agents or vaccines, who have had no cancer treatment for at least 24 months, and who have had no evaluable disease within 3 months of screening for this study may be eligible to participate.

Participants are randomly assigned to one of three study groups: Tai Chi, exercise training, or a waiting list. Individuals in the Tai Chi and exercise training groups participate in a supervised program for 1 hour 3 times a week for 12 weeks in the NIH Clinical Center's Rehabilitation Medicine department. Individuals assigned to the waiting list are followed for 12 weeks during the waiting period and are then assigned to either the Tai Chi or exercise program for another 12 weeks as described above.

At three time points during the study-before starting the program and after 6 weeks and 12 weeks of practicing the study intervention or being on the waiting list-participants undergo the following procedures:

Complete questionnaires regarding their quality of life and stress

Rehabilitation medicine evaluation, including the following:

* Questions about managing their daily activities, whether their skills have changed over time, what they may or may not have been able to do, or what they may have had to overcome as a result of their previous illness and the study program they have been practicing
* Measurements of strength and mobility
* Evaluation of overall physical fitness and endurance
* Blood tests to measure blood cell counts and cholesterol, lipid, hormone and mineral levels

DETAILED DESCRIPTION:
Diagnosis and treatment for cancer represent a major life-time stressor for any patient. While the diagnosis of a life-threatening illness is stressful, undergoing treatment for cancer including surgery, radiotherapy and chemotherapy result in stress to the patient. In addition, cancer treatment frequently is associated with fatigue, physical de-conditioning and metabolic abnormalities characteristic of the metabolic syndrome, leading to speculations that cancer therapy may render survivors more prone to developing metabolic syndrome and its sequelae, cardiovascular disease. In a recently conducted study we detected a high incidence of hyperlipidemia and increased body fat content, decreased aerobic performance and musculoskeletal functioning and a high frequency of parameters of psychological distress in long-term survivors of pediatric sarcoma. Based on these data and findings, it appears desirable to devise a program that would help cancer survivors not only to improve musculoskeletal functioning and aerobic performance, as a physical exercise program would offer, but in addition relieve psychological stress and enhance the well-being of cancer survivors after completion of treatment with multimodality therapy. Tai Chi Chuan (TCC) has been used in Asian culture for centuries to improve wellness, reduce stress, and to promote healing by improving the flow of Qi. While a number of studies have provided scientific support for these claims in different populations, a beneficial role for TCC in the management of cancer survivors has not been established.

This study aims to compare in a randomized, wait-list controlled design, the efficacy of TCC to an exercise program in improving aerobic exercise capacity and endurance, reducing stress and improving Quality of Life in adult survivors of malignant solid tumors.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this study, patients must meet the following criteria:

Diagnosis of solid cancer

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1

Age 18 - 65 years at time of study enrollment

Patients must be considered cancer survivors defined either as:

In the first continued remission from cancer after completion of initial therapy (i.e., No Evaluable Disease (NED) for greater than 2 years after successful completion of initial cancer therapy) or

In continued remission for greater than 5 years after completion of salvage therapy for disease recurrence

Must have completed cancer treatment regimen that includes chemotherapy, biologic agents (e.g. IL-2, interferon) or vaccines

Patients must have had no cancer treatment (e.g., chemotherapy, radiation therapy, cancer related surgery and/or immunotherapy) within the last 24 months

Patients must be free of recurrence at the time of evaluation (e.g., No Evaluable Disease (NED) by history and evaluation within the past 3 months)

Must be able to understand and sign consent.

EXCLUSION CRITERIA:

Diagnosis of hematologic malignancy

History of CAD/Angina or cardiomyopathy

History of CVA/stroke

Current clinical diagnosis of major depression

Prior or current practice of Tai Chi Chuan

Inability to perform and follow study intervention routine or study assessments/measures according to assessment of Principal Investigator, Rehabilitation Medicine Physician or TCC instructor (Dr. Adeline Ge).

Treatment with stimulants, antidepressants (for diagnosis of major depression), neuroleptics, betablockers or cardiac antiarrhythmics.

Current enrollment on or participation in a regular, structured exercise program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-10-26; Primary Completion 2007-07-31 (Actual); Study Completion 2011-02-25 (Actual)

PRIMARY OUTCOMES:
In adult solid cancer survivors, to determine that the TCC arm will have a larger reduction in psychological stress measured by the Perceived Stress Scale compared to the aerobic exercise and wait-list arms.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chernecky C. Temporal differences in coping, mood, and stress with chemotherapy. Cancer Nurs. 1999 Aug;22(4):266-76. doi: 10.1097/00002820-199908000-00003. PMID 10452203
- [Background] Hughes J. Emotional reactions to the diagnosis and treatment of early breast cancer. J Psychosom Res. 1982;26(2):277-83. doi: 10.1016/0022-3999(82)90047-2. PMID 7077559
- [Background] Sabbioni ME, Bovbjerg DH, Jacobsen PB, Manne SL, Redd WH. Treatment related psychological distress during adjuvant chemotherapy as a conditioned response. Ann Oncol. 1992 May;3(5):393-8. doi: 10.1093/oxfordjournals.annonc.a058214. PMID 1616894